CLINICAL TRIAL: NCT05028075
Title: Evaluating the Effectiveness of an Enhanced Digital Mental Health Care Delivery System
Brief Title: Health Care Workers and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 848844; 1R01MH127686-01 (NIH)
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Depressive Symptoms; Anxiety; Well-Being
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cobalt

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will complete baseline surveys at enrollment and then complete subsequent surveys (depression, anxiety, well-being, satisfaction with access to care, work productivity, hours of direct patient care, percent of time providing care for patients with COVID-19) at enrollment; 0 months, 6 months, and 9 months.
- Intervention (Experimental): Participants will complete baseline surveys at enrollment and then complete subsequent surveys (depression, anxiety, well-being, satisfaction with access to care, work productivity) at enrollment; 0 months and then again at 6 months and 9 months. The intervention group receives usual Cobalt plus: 1) monthly automated text messaging reminders and links to Cobalt resources 2) intermittent mental health assessments which triage individuals to an appointment based on their results.
  Interventions: Behavioral: Cobalt +

INTERVENTIONS:
Behavioral: Cobalt + — Participants will complete baseline surveys at enrollment and then complete subsequent surveys (depression, anxiety, well-being, satisfaction with access to care, work productivity) at enrollment; 0 months and then again at 6 months. The primary endpoint is assessed at 6 months. A secondary endpoint of persistence of effect is measured 3 months later-9 months post initiation. The intervention group receives usual Cobalt plus: 1) monthly automated text messaging reminders and links to Cobalt resources 2) intermittent mental health assessments which triage individuals to an appointment based on their results.
  Arms: Intervention

SUMMARY:
The purpose of this proposal is to deploy digital health interventions to bring timely, easily accessible resources and care to address the mental health and well-being needs of HCWs with direct patient care that are experiencing the impact of the COVID-19 pandemic and its economic, financial, and social sequelae at present and presumably for years to come. This proposal will evaluate the effectiveness of an enhanced digital mental health care delivery system (Cobalt), any differential effect by race and gender and, through qualitative interviews, how those interventions are perceived.

DETAILED DESCRIPTION:
The purpose of this proposal is to deploy digital health interventions to bring timely, easily accessible resources and care to address the mental health and well-being needs of HCWs with direct patient care that are experiencing the impact of the COVID-19 pandemic and its economic, financial, and social sequelae at present and presumably for years to come. This proposal will evaluate the effectiveness of an enhanced digital mental health care delivery system (Cobalt), any differential effect by race and gender and, through qualitative interviews, how those interventions are perceived. No Intervention: Usual Care, Participants will complete baseline surveys at enrollment and then complete subsequent surveys (depression, anxiety, well-being, satisfaction with access to care, work productivity, hours of direct patient care, percent of time providing care for patients with COVID-19) at enrollment; 0 months, 6 months, and 9 months. Behavioral: Cobalt +: Participants will complete baseline surveys at enrollment and then complete subsequent surveys (depression, anxiety, well-being, satisfaction with access to care, work productivity) at enrollment; 0 months and then again at 6 months. The primary endpoint is assessed at 6 months. A secondary endpoint of persistence of effect is measured 3 months later-9 months post initiation. The intervention group receives usual Cobalt plus: 1) monthly automated text messaging reminders and links to Cobalt resources 2) intermittent mental health assessments which triage individuals to an appointment based on their results.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Regular, daily access to an smartphone
3. Able to communicate fluently in English
4. Work at least 4 hours per week in either a hospital or outpatient based setting. This includes health care workers like physicians, nurses, certified nursing assistants, lab technicians, radiology technicians, physical therapist, occupational therapist, pharmacists, pharmacy technicians, patient registration staff, receptionists/patient intake coordinators, environmental and food service personnel approximately 4 hours/week. This averages 192 hours/ 48 weeks in a year) in the study time frame.

Exclusion Criteria:

1. Not aged 18 years or older
2. Does not have regular, daily access to a smartphone
3. Unable to communicate fluently in English
4. Does not work at least 4 hours per week in either a hospital or outpatient based setting.
5. Not willing to sign the informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Southwick L, Gonzales R, Bellini L, Asch DA, Mitra N, Balachandran M, Wolk CB, Becker-Haimes EM, Kishton R, Beck S, Merchant RM, Agarwal AK. Proactively Delivered Digital Mental Health Support for Health Care Workers: Usability and Acceptability Evaluation. JMIR Form Res. 2025 Dec 9;9:e74086. doi: 10.2196/74086. PMID 41364911
- [Derived] Agarwal AK, Southwick L, Gonzales RE, Bellini LM, Asch DA, Shea JA, Mitra N, Yang L, Josephs M, Kopinksy M, Kishton R, Balachandran M, Benjamin Wolk C, Becker-Haimes EM, Merchant RM. Digital Engagement Strategy and Health Care Worker Mental Health: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2410994. doi: 10.1001/jamanetworkopen.2024.10994. PMID 38787562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 633 | 642
Completed | 509 | 462
Not Completed | 124 | 180

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 633 | 642 | 1275
Age, Continuous [Mean (Standard Deviation); unit: age] | 38.6 (11.1) | 38.6 (10.6) | 38.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529 | 534 | 1063
  Male | 104 | 108 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 39 | 77
  Not Hispanic or Latino | 595 | 603 | 1198
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 54 | 55 | 109
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 160 | 160 | 320
  White | 394 | 399 | 793
  More than one race | 17 | 21 | 38
  Unknown or Not Reported | 0 | 0 | 0
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] | 5.71 (4.74) | 5.92 (5.19) | 5.81 (4.97)
GAD-7 [Mean (Standard Deviation); unit: units on a scale] | 5.79 (4.77) | 6.03 (4.88) | 5.91 (4.83)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Score Change
Description: Patient health questionnaire-9 (PHQ-9) (Kroenke, Spitzer, & Williams, 2001) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. PHQ-9 is brief and useful in clinical practice. The PHQ-9 is completed by the patient in minutes and is rapidly scored by the clinician. The PHQ-9 is a freely available mood-rating questionnaire consisting of nine questions mirroring DSM-IV depression diagnostic criteria. The PHQ-9 has shown diagnostic validity in a study of 3,000 adult patients. Each item is rated on a scale of 0 to 3, giving a maximum score of 24. Cut-off scores are used to label depression severity as: 0 to 4, minimal depression; 5 to 9, mild depression; 10 to 14, moderate depression; 15 to 19, moderately severe depression; 20 to 24, severe depression.
Time Frame: 6 months and baseline measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 508 | 462
units on a scale | 5.29 (4.93) | 4.65 (4.73)

2. Primary Outcome: Anxiety Symptoms Score Change
Description: GAD-7 is a 7-item anxiety scale. It has good reliability, as well as criterion, construct, factorial, and procedural validity. Each item is rated according to the frequency of the described problem. The responses are scored as follows: 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day with a maximum score of 21 Scores are interpreted as 5 to 9, mild anxiety; 10 to 14, moderate anxiety; and 15 and above, severe anxiety. The GAD-7 showed good reliability and criterion, construct, factorial, and procedural validity in a study carried out in 15 primary care clinics. The GAD-7 is a valid and efficient tool for screening for GAD and assessing its severity in clinical practice and research.
Time Frame: 6 months and baseline measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 509 | 462
units on a scale | 5.54 (4.81) | 5.00 (4.90)

3. Secondary Outcome: Well-being Score Change
Description: The Well-being index (WBI) is a nine-question survey validated for use in Health Care Worker populations and considered important to health systems in managing the well-being of their workforce. The original 7-item WBI items are answered ''yes/no'' with 1 point assigned for each ''yes'' response. A total score (0 - 7) is calculated by adding the number of ''yes'' responses. A higher score indicative of worse well-being.
Time Frame: 6 months and baseline measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 528 | 484
units on a scale | 2.24 (2.30) | 2.05 (2.34)

4. Secondary Outcome: Work Productivity Score Change
Description: To evaluate work productivity, we will use Lam Employment Absence and Productivity Scale, or LEAPS. It is a 10-item, self-rated scale that takes only 3 to 5 minutes for the patient to complete. It is simple and easy to use. The items were chosen based on the symptoms that have the most impact on work productivity and the most common productivity problems experienced by patients with depression. The LEAPS was recently validated in a sample of 234 consecutive working patients meeting DSM-IV criteria for MDD attending a mood disorders outpatient clinic. Each question has 5 choices ranging from none of the time, some of the time, half of the time, most of the time, and all of the time. Each choice is scored from 0 to 4. The total score is summing the 7 questions, the total score can range from 0 to 28. A lower score represents no to minimal work impairment while a higher score represents severe work impairment.
Time Frame: 6 months and baseline measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 517 | 473
units on a scale | 5.25 (4.08) | 4.94 (4.34)

5. Secondary Outcome: Psychological Well-being Score Change
Description: The 5-item World Health Organization Well- Being Index (WHO-5) is among the most widely used questionnaires assessing subjective psychological well-being. The five questions are scored from 0 to 5. The raw score is calculated by totaling the figures of the five answers.The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life. To obtain a percentage score, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Time Frame: 6 months and baseline measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 508 | 461
units on a scale | 13.88 (5.23) | 14.15 (5.43)

ADVERSE EVENTS:
Time Frame: Adverse events were collected the duration of the randomized controlled trial (9-months).
Description: The number of participants at risk for Serious Adverse Events, All-Cause Mortality, Adverse is zero.
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/633 | 0/642
Serious Adverse Events (participants affected / at risk) | 0/633 | 0/642
Other Adverse Events (participants affected / at risk) | 0/633 | 0/642

LIMITATIONS AND CAVEATS:
Participants were from a single, large, urban health system and needed daily access to a smartphone. Selection and non-responder bias may be present. Given the stigma with accessing mental health care, this study did not integrate mental health records or treatments received but rather gathered self-reported data from participants and data on appointments made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT05028075/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT05028075/ICF_002.pdf